CLINICAL TRIAL: NCT01258062
Title: Phase 1, Double Blind, Randomized, Placebo Controlled Study to Assess Safety and Immunogenicity of an Inactivated H5N1 Influenza Vaccine Administered in GelVac Nasal Powder to Healthy Young Adults.
Brief Title: Study to Assess Safety of an Inactivated H5N1 Influenza Vaccine Administered in GelVac Nasal Powder to Healthy Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-GEL-NT/001
Record Dates: First submitted 2010-12-06; First posted 2010-12-10 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Phase 1 Safety Study of GelVac Nasal Powder H5N1 Influenza Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- of GelVac™ nasal powder H5N1 influenza vaccine. (Experimental)
  Interventions: Drug: GelVac™ nasal powder H5N1 influenza vaccine.
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GelVac™ nasal powder H5N1 influenza vaccine. — subjects will be randomized to either 30 µg of Inactivated H5N1 Influenza Vaccine Administered in GelVac™ Nasal Powder given as two doses of 15 μg in one nostril or placebo vaccine given as two doses administered in GelVac™ Nasal Powder in one nostril
  Arms: of GelVac™ nasal powder H5N1 influenza vaccine.
Drug: Placebo — subjects will be randomized to either 30 µg of Inactivated H5N1 Influenza Vaccine Administered in GelVac™ Nasal Powder given as two doses of 15 μg in one nostril or placebo vaccine given as two doses administered in GelVac™ Nasal Powder in one nostril
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo controlled, safety and immunogenicity study of GelVac™ nasal powder H5N1 influenza vaccine. Healthy male and female subjects between 18 and 49 years of age who are eligible for study participation will be enrolled in the trial. It is expected that 10 subjects will be screened to obtain 7 subjects who will be eligible for study participation.

The primary objective is to determine the frequency and severity of local and systemic adverse events of vaccine.

The secondary objective is to assess the immunogenicity of the vaccine based on geometric mean titers (GMT) of serum HAI, serum neutralizing, and nasal wash IgA antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. able to read and sign Informed Consent Form (ICF).
2. male or female > 18 and < 49 years of age at the time the ICF is signed.
3. generally healthy, as determined by medical history and clinical assessment.
4. able to attend all scheduled visits and to comply with all trial procedures.
5. if female of child-bearing potential, use of an acceptable method of contraception or abstinence for at least 4 weeks prior to the first vaccination through at least four weeks after the second vaccination. Acceptable methods are hormonal birth control or a barrier method with spermicide.
6. if female, post menopausal (no menstrual period within the last 12 months), surgically sterile (hysterectomy or tubal ligation), or have a negative urine pregnancy test within 24 hours prior to the time of vaccination.

Exclusion Criteria:

1. has a known allergy to fruits (e.g., apples, oranges) or pectin and/or pectin by-products (including jams or jellies).
2. has a known allergy to dairy/milk products/lactose.
3. is breast-feeding or pregnant or planning on becoming pregnant within 1 month of vaccination.
4. has a history of a chronic viral infection (i.e.; Shingles, Herpes Zoster, HIV).
5. has a history of severe allergic reaction following influenza vaccination, systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing the same substances.
6. has a history of demyelinating disease (esp. Guillian-Barre Syndrome).
7. history of Bell's Palsy.
8. immunosuppression as a result of underlying illness or treatment.
9. use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) within 1 month prior to vaccination.
10. use of other immunosuppressive or cytotoxic drugs or radiation therapy within six months prior to vaccination.
11. use of OTC or other 'herbal' immune suppressant or stimulants within the 6 months prior to vaccination.
12. active neoplastic disease or history of any hematologic malignancy in the past 5 years (except localized skin or prostate cancer that is stable in the absence of therapy).
13. acute or chronic condition that (in the opinion of the Investigator) would render vaccination unsafe or would interfere with the evaluation of responses including, but not limited to the following: known chronic liver disease, significant renal disease, oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV, unstable or progressive neurologic disorder, insulin-treated diabetes mellitus, and asthma.
14. use of experimental vaccines within 6 months prior to study entry, or expected use of experimental vaccines during the entire study period after inoculation with study vaccine.
15. participation in another clinical trial 30 days prior to study entry.
16. use of experimental devices or participation in a medical procedure trial within the month prior to study entry, or expected use of experimental devices or participation in a medical procedure trial during the entire study period.
17. receipt of immunoglobulin or other blood product within 3 months prior to enrollment.
18. receipt of other licensed vaccines within the preceding 6 months or expected to receive a licensed vaccine within 28 days following last trial vaccination.
19. subject is enrolled in a conflicting clinical trial.
20. any disorder or therapy contraindicating influenza vaccination.
21. Have a clinically significant structural abnormality of the nasopharynx (e.g., obvious deviation that obstructs airflow in either nostril), as determined by the investigator
22. acute respiratory disease at the time of enrollment.
23. febrile illness with temperature greater than or equal to 38 degrees Celsius (100.4 degrees F) within 72 hours prior to enrollment.
24. receipt of allergy shots within the preceding 7 days or expected to receive allergy shots within 7 days following vaccination.
25. any condition that, in the opinion of the investigator, would pose a health risk to the participant.
26. presence of any active disease or condition at the administration site that, in the opinion of the Investigator, would impact vaccine delivery or assessment of vaccination site.
27. history of drug abuse or alcohol abuse in the five years prior to enrollment. Subject who abuses alcohol or other drugs of abuse.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the frequency of adverse events of the vaccine. | up to 26 weeks

SECONDARY OUTCOMES:
The secondary objective is to assess the immunogenicity of the vaccine based on geometric mean titers (GMT) of serum HAI. | up to 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Research Network, LLC, Gainesville, Florida, United States